CLINICAL TRIAL: NCT05043584
Title: Autofluorescence-guided Thyroid Surgery: Impact on Parathyroid Preservation and Hypoparathyroidism
Brief Title: Near-infrared Autofluorescence (NIRAF)-Guided Total Thyroidectomy: Impact in Low-volume, Non-parathyroid Institutions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regional Hospital West Jutland (Other)
Collaborators: Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Responsible Party: Principal Investigator, Ali Abood, Principal Investigator, Regional Hospital West Jutland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Autofluorescence1.0
Record Dates: First submitted 2021-09-05; First posted 2021-09-14 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Autofluorescence; Thyroidectomy; Hypoparathyroidism; Hypocalcemia
MeSH Terms: conditions — Hypoparathyroidism; Hypocalcemia

STUDY DESIGN:
Intervention Model Description: Prospective cohort study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- (A): NIRAF-assisted surgery (Experimental): Patients undergoing NIRAF-assisted total thyroidectomy
  Interventions: Device: Fluobeam LX, Fluoptics, Grenoble, France

INTERVENTIONS:
Device: Fluobeam LX, Fluoptics, Grenoble, France — See arm description

SUMMARY:
Hypoparathyroidism is the most frequent complication in total thyroidectomy. The use of near-infrared autofluorescence (NIRAF) intraoperatively, seems to reduce the rate of transient hypoparathyroidism. Unfortunately, no effect on permanent hypoparathyroidism has been shown.

In order to cover every aspect of the impact of NIRAF in thyroid surgery, an evaluation in low-volume, non-parathyroid institutions is needed. This is the overall aim of our current studies. The objective of this specific study is to evaluate the impact of NIRAF on immediate, transient and permanent hypoparathyroidism following total thyroidectomy in low-volume, non-parathyroid institutions.

DETAILED DESCRIPTION:
Patients referred for total thyroidectomy will undergo NIRAF-assisted surgery (Fluobeam LX) at two low-volume ENT-departments with no experience in parathyroid surgery.

PTH and ionized calcium will be assessed preoperatively, on postoperative day 1 (POD1) and minimum two months following surgery. Patients who still fulfill the criteria for hypoparathyroidism at that point will be followed until one year following surgery. The rates of immediate, transient and permanent hypoparathyroidism will be assessed and compared to a historic cohort.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for total thyroidectomy
* Age > 18
* Able to understand patient information
* Able to give informed consent

Exclusion Criteria:

* Previous thyroid surgery
* Need for accelerated surgery
* Insufficient biochemical profile

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Rate of hypoparathyroidism | Will be assessed on postoperative day one, minimum two months and one year following surgery.

SECONDARY OUTCOMES:
Parathyroid gland identification rate | Will be assessed at the time of surgery
Parathyroid autotransplantation rate | Will be assessed at the time of surgery
Rate of inadvertently excised parathyroid glands | Will be assessed 1 month following surgery

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Department of Otorhinolaryngology, Hospital South West Jutland, Esbjerg
  - Department of Otorhinolaryngology, Regional Hospital West Jutland, Holstebro

IPD SHARING:
Plan to Share IPD: No